CLINICAL TRIAL: NCT06947447
Title: WatchPAT SpO2 Validation Study
Status: Completed | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Collaborators: Element Materials Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: PR# 2024-598
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Arterial Oxygen Saturation; Oxygen Saturation; WatchPAT; SpO2 sensor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- WatchPAT SpO2: Simultaneous data collection will be set up for the reference(s) and the device under test. The participants will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels. The WatchPAT will be placed on the finger(s) of both hands following the instructions for use.
  Each participant test is expected to take approximately 1.5 to 2 hours.
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention — Device

SUMMARY:
Validate the SpO2 accuracy of the WatchPAT compared to arterial blood CO-Oximetry

DETAILED DESCRIPTION:
The goal of this comparative, single-center, non-randomized study is to validate the SpO2 accuracy performance of the WatchPAT SpO2 sensor over the range of 70-100% SaO2 during non-motion conditions assessed by CO-Oximetry in 24 healthy male and female participants of any race, ranging in pigmentation from light to dark, aged 18-50 years old. The participants will have an arterial catheter placed in the radial artery to allow for simultaneous blood samples during stable plateaus of induced hypoxic levels, while an investigational device will be placed on the fingers of both hands.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have the ability to understand and provide written informed consent.
* Participant is adult 18-50 years of age.
* Participant must be willing and able to comply with study procedures and duration.
* Participant is a non-smoker or who has not smoked within 2 days prior to the study.
* Male or female of any race.

Exclusion Criteria:

* Participant is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation (i.e., Raynaud's Syndrome), injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoos in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the sites utilized.)
* Females who are pregnant, who are trying to get pregnant, (confirmed by positive urine pregnancy test unless the participant is known to be not of child-bearing potential)
* Participants who have smoked in the last 2 days or participants who have refrained, for at least 48 hours, with COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Participants with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery,
  * emphysema, COPD, lung disease
  * Recent COVID with hospitalization
* Participants with self-reported heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * high blood pressure: systolic >140 mmHg or diastolic >90 mmHg on 3 consecutive readings (reviewed during health screen)
  * have had cardiovascular surgery, except successful minor surgery without clinical symptoms (i.e., PFO, PDA)
  * chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
  * implantable active medical device such as pacemaker or automatic defibrillator
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent symptomatic head injury (within the last 2 months),
  * Cancer requiring chemotherapy, radiation, or current treatment.
* Participants with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
  * Sickle Cell Trait or Disease
* Participants with severe contact allergies to standard adhesives, latex, silicone or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Participants with severe allergies to iodine (only applicable if iodine is used)
* Participants with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocaine),
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio <0.4)
* Unwillingness or inability to remove colored nail polish or non-clear artificial nails from test digits.
* Surgical hardware in pathway of Device Under Test
* Other known health conditions should be considered upon disclosure in health assessment form.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 healthy male and female participants of any race, ranging in pigmentation from light to dark, aged 18-50 years old
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy | April-May 2025
  WatchPAT SpO2 accuracy performance over the range of 70-100% SaO2 during non-motion conditions assessed by CO-Oximetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No